CLINICAL TRIAL: NCT02732925
Title: Multiple Myeloma Spinal Disease Study; A Multi-centre, Prospective, Single Blinded, Randomized, Controlled Study to Compare Conservative Management Alone Vs. Balloon Kyphoplasty With the Treatment of VCFs in Patients With Multiple Myeloma
Brief Title: To Compare Conservative Management Vs. Balloon Kyphoplasty in the Treatment of VCFs in Patients With Multiple Myeloma
Acronym: MELODY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with recruitment due to change in referral rates.
Sponsor: Royal National Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Iva Hauptmannova, Head of Research Innovation Centre, Royal National Orthopaedic Hospital NHS Trust
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RNOH - Melody Study
Record Dates: First submitted 2014-11-03; First posted 2016-04-11 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Multiple Myeloma
Keywords: Vertebral Compression Fracture; Balloon Kyphoplasty; Conservative treatment; Sham procedure; VCFs; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Sham Procedure (Sham Comparator): Sham Procedure & Conservative Treatment
  Subjects will be blinded and randomised to Arm 1 and will undergo a general anaesthetic and undergo a sham procedure. They will also be treated under conservative management alone.
  Below is a list of the conservative management they will be managed by their Doctor:
  1. Bisphosphonates
  2. Pain relief
  3. Systemic chemotherapy for Myeloma disease
  4. Bed rest
  5. Radiotherapy
  6. Physiotherapy
  This is a non interventional as conservative treatment (standard of care for multiple myeloma patients) is used.
  Interventions: Procedure: Conservative Management
- Arm 2 - Balloon Kyphoplasty (Active Comparator): Balloon Kyphoplasty & Conservative Treatment - Interventional Arm
  Subjects will be blinded and randomised to Arm 2 (balloon kyphoplasty) and will undergo a general anaesthetic and undergo a balloon kyphoplasty surgical procedure. They will also be treated with conservative management.
  Below is a list of the conservative management they will be managed by their Doctor:
  1. Bisphosphonates
  2. Pain relief
  3. Systemic chemotherapy for Myeloma disease
  4. Bed rest
  5. Radiotherapy
  6. Physiotherapy
  This is a interventional arm (balloon kyphoplasty procedure) and the patient will receive conservative treatment (standard of multiple myeloma patients) is used.
  Interventions: Device: Arm 2 Balloon Kyphoplasty; Procedure: Conservative Management

INTERVENTIONS:
Device: Arm 2 Balloon Kyphoplasty — Arm 2 Balloon Kyphoplasty (Medtronic LCC) and Conservative Treatment
  Subjects will be blinded and randomised to Arm 2 and will undergo a general anaesthetic and undergo a balloon kyphoplasty surgical procedure. They will also be treated with conservative management.
  Below is a list of the conservative management they will be managed by their Doctor:
  1. Bisphosphonates
  2. Pain relief
  3. Systemic chemotherapy for Myeloma disease
  4. Bed rest
  5. Radiotherapy
  6. Physiotherapy
  Arms: Arm 2 - Balloon Kyphoplasty
Procedure: Conservative Management — Patients recruited to Arm 1 and Arm 2 will undergo conservative management for Multiple Myeloma recommended by their Consultant Hematologist.
  * Concomitant treatment with bisphosphonates
  * Pain relief as required
  * Systemic chemotherapy for Myeloma disease
  * Bed rest
  * Radiotherapy
  * Physiotherapy

SUMMARY:
The purpose of this study is to determine whether surgical treatment, balloon kyphoplasty is more effective compared to conservative treatment alone (sham procedure) when assessing clinical, translational, radiological & patient outcomes in patients with multiple myeloma.

Subjects will be recruited to the study if they have VAS score ≥ 6 and has given informed consent to participate in the Melody Study will be randomised to Arm 1 Sham Procedure and Conservative treatment or Arm 2 Balloon Kyphoplasty and Conservative treatment. Subjects recruited to Arm 1 (Sham Procedure and Conservative treatment) can cross over into Arm 2 (Balloon Kyphoplasty and Conservative Treatment) if they have a VAS score ≥ 6 between 8-12 weeks.

DETAILED DESCRIPTION:
Multiple myeloma (MM) accounts for 10% of the malignant haematological diseases and approximately 1% of all cancer-related deaths in Western countries. MM is characterised by the accumulation of malignant plasma cells in the bone marrow leading to impaired haematopoiesis and the highest incidence of bone involvement among the malignant diseases. MM bone disease is the result of increased destruction of bone that cannot be compensated for by new bone formation. Approximately 80% of patients with MM develop skeletal complications including bone pain, hypercalcemia, osteoporosis, osteolytic lesions and pathologic fractures. Vertebral fractures may be associated with spinal cord compression and neurological complications requiring surgery and/or radiotherapy. Osteolytic bone destruction is the most debilitating manifestation of MM, has a severe impact on patients' quality of life and is responsible for increased morbidity and mortality. Furthermore, bone resorption activity has been shown to be an independent risk factor for overall survival in patients with symptomatic MM. Moreover, myeloma-associated lytic bone lesions do not repair, even in patients who are disease free for years.

More than 50% of patients develop vertebral compression fractures (VCFs) either by the time of diagnosis or during the course of the diagnosed disease. These fractures can compromise the spinal cord and patients' height and stature, cause angulation of the spine, increasing sternum pressure, eventually resulting in sternal fractures and compromising the pulmonary capacity. 9% loss in predicted forced vital capacity is associated with each vertebral fracture. Deformity, Insomnia, depression, substantial physical, functional and psychological impairment and ultimately disability can be the result of severe vertebral compression fractures poorly managed at presentation.

Management of spinal MM bone disease

1. Bisphosphonates he use of bisphosphonates, which inhibit bone reabsorption, for the treatment of MM bone disease has led to an improvement in the quality of life for patients with MM.
2. Conservative (non-surgical) management (this is standard of care management for patients with multiple myeloma)

   1. Pain relief
   2. Systemic chemotherapy for Myeloma disease
   3. Bed rest
   4. Radiotherapy
   5. Physiotherapy
3. Standard surgical procedures

A. Open surgical decompression Anterior or posterior decompression and stabilisation through internal fixation hardware and bone grafting (in <0.5% with gross spinal deformity or neurologic impairment). Higher morbidity and mortality in MM patients because of comorbid conditions related to age, disease associated end-organ damage and immunosuppression B. Minimally invasive - Cement Augmentation

1. Percutaneous Vertebroplasty
2. Percutaneous Kyphoplasty (i.e. Balloon Kyphoplasty)

COST BURDEN, HEALTH ECONOMIC IMPACT AND COST UTILITY ANALYSIS There is little evidence on differences across health systems in choice and outcome of multiple myeloma being treated with conservative treatment, chemotherapy and spinal surgery are three of many treatment options for managing multiple myeloma. The true cost associated with current therapies in addition to supportive care, is significant and poses a tremendous financial burden to both patient and health care providers.

There is therefore a need to begin to systematically optimise the guidance for treatment for this subgroup of patients especially when comparing the two treatment arms in this study, conservative treatment alone versus surgical treatment, balloon kyphoplasty.

This study will determine the cost burden, health economic impact and cost utility analysis by combining the quality of life measurements, the cost analysis will allow a calculation of the relative cost-effectiveness of conservative treatment standard of care versus standard of care plus balloon kyphoplasty.17

RATIONALE FOR CURRENT STUDY

Osteolytic lesions of vertebral bodies are frequent problems in multiple myeloma patients predisposing to severe pain, vertebral fractures and consequent neurological complications.Open surgical procedures to stabilise or correct deformed vertebral bodies are associated with major complications in this group of immunocompromised patients. In addition, open procedures are often not possible, due to a severely impaired strength of the bone tissue, which does not allow the safe application of screws and plates. As a result the standard management to reduce the local pain secondary to vertebral compression fracture has for many years been with pain relief, radiotherapy and the other elements of conservative management listed above. The development of minimally invasive procedures such as kyphoplasty and vertebroplasty has been demonstrated to be an additional effective treatment option to improve mobility and quality of life and to reduce pain.

Percutaneous vertebroplasty involves the injection of acrylic bone cement into the vertebral body in order to relieve pain and/or stabilise the fractured vertebrae and in some cases, restore vertebral height.

Percutaneous Kyphoplasty (or Balloon Kyphoplasty) is performed by inserting a balloon-like device (inflatable bone tamp) through a channel created by a hand drill in the fractured vertebrae. The tamp is positioned and inserted into the vertebral body. The balloon is then inflated slowly until normal height of the vertebral body is restored or the balloon reaches its maximum volume. The procedure is intended to restore vertebral height and correct kyphosis. It may also help to improve pulmonary and gastrointestinal function and reduce the likelihood of subsequent vertebral compression fractures. The inflation of the balloon tamp creates a cavity in the vertebral body so that when the bone tamp is withdrawn, bone cement can be injected into the cavity at a lower pressure, potentially reducing the risk of cement leakage. The cement increases the strength of the vertebra and is intended to provide pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤80 years old
* Diagnosis of Multiple Myeloma
* Confirmed acute (MRI, a detectable low signal T1 ± oedema) painful vertebral compression fracture(s) VAS score is ≥6
* The patient is able to read and understand the Patient Information Sheet and study procedures
* The patient is able and willing to give written informed consent

Exclusion Criteria:

* Contraindications to anaesthesia
* Cord Compression or large epidural mass necessitating conservative management before balloon kyphoplasty
* Pain unrelated to vertebral collapse
* Infection at the site
* Presence of overt instability as judged by the principle investigator
* Known pregnancy at time of screening
* Severe Cardiopulmonary insufficiency
* Osteoblastic lesions
* Any co-morbidity, (e.g., diabetes, heart condition, obesity, psychiatric illness) which, in the opinion of the investigator, is of a severe enough nature to; interfere with the patient's ability to complete the study assessments; or present an unacceptable risk to the patient's safety to undergo study treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
the effect of sham procedure & conservative management alone (arm 1) versus balloon kyphoplasty (arm 2) on patient reported pain scores as assessed by VAS (at week 4) | At week 4

SECONDARY OUTCOMES:
the effect of conservative management alone versus balloon kyphoplasty on patient reported pain scores as assessed by VAS (at weeks 1, 8, 12, 16, 26, year 1 and year 2) | At week 1, 8, 12, 26, year 1 and year 2
the pain relief requirements of conservative management alone versus balloon kyphoplasty using a daily pain diary (capturing usage of pain relief by type) | At week 1, 8, 12, 26, year 1 and year 2
the effect of conservative management alone versus balloon kyphoplasty on patient reported Quality Of Life outcomes | At week 1, 8, 12, 26, year 1 and year 2
procedure related complications of conservative management alone versus balloon kyphoplasty | At week 1, 8, 12, 26, year 1 and year 2
  recording of any adverse events
the cost utility of the conservative management alone versus the balloon kyphoplasty | at 2 years
  Data collected for all intervention groups from the study will be assessed to compare the overall cost of care for conservative management vs. kyphoplasty

CONTACTS AND LOCATIONS:
Overall Officials: Chara Kyriakou, MD PhD, Principal Investigator — RNOH; Sean Molloy, FRCS MSc, Principal Investigator — RNOH
Locations (1):
- Royal National Orthopaedic NHS Trust, Brockley Hill, Stanmore, UK, United Kingdom